CLINICAL TRIAL: NCT06756503
Title: Prevalence and Clinical Characteristics of Exocrine Pancreatic Insufficiency in Patients With Functional Dyspepsia
Brief Title: Exocrine Pancreatic Insufficiency and Functional Dyspepsia
Status: Not yet recruiting | Type: Observational
Sponsor: Maria Marta Piskorz (Other)
Responsible Party: Sponsor-Investigator, Maria Marta Piskorz, Principal Investigator, Hospital de Clinicas José de San Martín
Organization: Hospital de Clinicas José de San Martín (Other)
Other Study IDs: HCJSM-10-2024
Record Dates: First submitted 2024-10-22; First posted 2025-01-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Exocrine Pancreatic Insufficiency; Dyspepsia
Keywords: Exocrine pancreatic insufficiency; Functional dyspepsia; Fecal elastase
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Dyspepsia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood extraction Fecal sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: fecal elastase — To investigate exocrine pancreatic insufficiency (EPI), all patients will be asked to provide a stool sample for fecal elastase (Fel-1) analysis. Participants will be instructed to collect their stool sample in a sterile, disposable plastic container and submit it to the Gastroenterology Chemistry Laboratory (Litwin Laboratory) for processing and analysis. Based on previously published reports, samples will be refrigerated at 4-8 °C for no more than 48 hours. The concentration of Fel-1 in all samples will be measured using a commercially available enzyme-linked immunosorbent assay (ELISA) kit (ScheBo-Pancreatic Elastase 1™, Giessen, Germany), with fecal elastase extracted and analyzed according to the manufacturer's instructions.
Diagnostic Test: Serum cytokines — Cytokines will be quantified using the Bio-Plex Pro™ Human Cytokine 27-plex commercial kit (Bio-Rad Laboratories, USA) following the kit instructions.

SUMMARY:
The goal of this observational study is to learn about the prevalence of exocrine pancreatic insufficiency in patients with functional dyspepsia .

. The main questions it aims to answer are: What is the prevalence of exocrine pancreatic insufficiency (EPI) in patients with functional dyspepsia? Wich are the clinical characteristics associated with (EPI) in patients with functional dyspepsia? Patients diagnosed with functional dyspepsia will undergo an evaluation of clinical symptoms and fecal elastase determination. In those with fecal elastase levels below 100 µg/g, an endoscopic ultrasound and other assessments will be performed to define the cause of exocrine pancreatic insufficiency (EPI).

DETAILED DESCRIPTION:
Functional dyspepsia and exocrine pancreatic insufficiency (EPI) represent two gastrointestinal disorders that can occur concomitantly. Functional dyspepsia involves chronic digestive symptoms without identifiable organic causes, while EPI refers to insufficient pancreatic enzyme production for adequate digestion.

Functional dyspepsia is prevalent in the general population, with estimates ranging from 10% to 30% based on various studies. Defined by Rome IV criteria, functional dyspepsia includes epigastric pain, early satiety, or postprandial bloating in the absence of organic conditions. EPI may occur more frequently in individuals with functional dyspepsia. Small studies have identified EPI as a potential mechanism contributing to symptoms. Dyspepsia has been identified as an independent predictor of EPI in research exploring this condition within irritable bowel syndrome.

Recent findings suggest a possible association between EPI and functional dyspepsia. Research by Tahtaci et al. (2018) evaluated EPI in a cohort with functional dyspepsia, revealing that approximately 15% of these patients met criteria for EPI. These findings underscore the importance of evaluating EPI in cases of persistent symptoms unresponsive to conventional treatment. Early identification of EPI may enhance therapeutic management and improve quality of life in this population.

Further studies remain necessary to elucidate the relationship between functional dyspepsia and EPI, establish precise diagnostic criteria, and optimize treatment strategies.

This study adopts a prospective, cross-sectional, and analytical design. A total of 65 patients with functional dyspepsia will undergo assessments including:

* Symptom severity questionnaires addressing depression, anxiety, somatization, and stress.
* Pancreatic Exocrine Insufficiency Questionnaire (PEI-Q).
* Alcohol and tobacco use (anticipated to correlate with higher prevalence of chronic pancreatitis).
* Measurements of weight, height, and abdominal circumference.
* Fecal elastase-1 (Fel-1) testing.
* Serum analysis of pro- and anti-inflammatory cytokines.
* Hydrogen and methane breath testing for small intestinal bacterial overgrowth (SIBO).

EPI will be diagnosed based on fecal elastase-1 concentrations <100 µg/g or values between 100 and 200 µg/g in conjunction with abnormalities in additional pancreatic pathology tests, including serum albumin, vitamin E, vitamin D, vitamin A, folic acid, iron, transferrin, calcium, magnesium, or evidence of malnutrition from anthropometric measurements by a nutritionist. Fecal elastase values ≥200 µg/g will be considered normal.

Patients with fecal elastase values below 200 will undergo additional testing, including:

- Proteinogram, vitamin E, vitamin D, vitamin A, vitamin K, folic acid, B12, calcium, magnesium, zinc, iron profile, and nutritional assessment with anthropometry.

For patients diagnosed with EPI, additional evaluations will include:

- IgG4, alpha-1 antitrypsin, and endoscopic ultrasound.

Based on these parameters, patients will be categorized into EPI and non-EPI groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age diagnosed with functional dyspepsia based on Rome IV criteria, who have been excluded for organic, metabolic, and medication-related causes (NSAIDs), and who test negative for H. pylori.

Exclusion Criteria:

* Pregnancy or lactation
* Organic diseases of the digestive tract (celiac disease, inflammatory bowel diseases, neoplasms, positive for H. pylori)
* Uncontrolled systemic diseases (diabetes mellitus, hypo- or hyperthyroidism, cancer, etc.)
* Lack of informed consent
* Severe psychiatric disorders, defined based on the DSM-5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age diagnosed with functional dyspepsia based on Rome IV criteria, who have been excluded for organic, metabolic, and medication-related causes (NSAIDs), and who test negative for H. pylori.
  The Rome IV criteria for functional dyspepsia include the presence of one or more of the following symptoms: bothersome postprandial fullness, early satiation, epigastric pain, or epigastric burning, occurring at least once a week in the last three months with symptom onset at least six months prior to diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
EPI prevalence | At baseline
  Determine the prevalence of exocrine pancreatic insufficiency (EPI) in patients with functional dyspepsia

SECONDARY OUTCOMES:
Groups comparison (EPI vs non EPI) | At baseline
  Define the clinical characteristics of patients group.
Factors associated with exocrine pancreatic insufficiency | At baseline
  To investigate the factors associated with EPI in patients with dysfunctional dyspepsia

IPD SHARING:
Plan to Share IPD: No
The data sets, including the redacted study protocol, redacted statistical analysis plan, and individual participant data supporting the results reported in this article, will be made available within 3 months from initial request to researchers who provide a methodologically sound proposal. The data will be provided after its de-identification, in compliance with applicable privacy laws, data protection, and requirements for consent and anonymization.

REFERENCES:
- [Result] Dominguez-Munoz JE. Diagnosis and treatment of pancreatic exocrine insufficiency. Curr Opin Gastroenterol. 2018 Sep;34(5):349-354. doi: 10.1097/MOG.0000000000000459. PMID 29889111
- [Result] Johnson CD, Williamson N, Janssen-van Solingen G, Arbuckle R, Johnson C, Simpson S, Staab D, Dominguez-Munoz E, Levy P, Connett G, Lerch MM. Psychometric evaluation of a patient-reported outcome measure in pancreatic exocrine insufficiency (PEI). Pancreatology. 2019 Jan;19(1):182-190. doi: 10.1016/j.pan.2018.11.013. Epub 2018 Nov 27. PMID 30528109
- [Result] Phillips ME, Hopper AD, Leeds JS, Roberts KJ, McGeeney L, Duggan SN, Kumar R. Consensus for the management of pancreatic exocrine insufficiency: UK practical guidelines. BMJ Open Gastroenterol. 2021 Jun;8(1):e000643. doi: 10.1136/bmjgast-2021-000643. PMID 34140324
- [Result] Tack J, Talley NJ, Camilleri M, Holtmann G, Hu P, Malagelada JR, Stanghellini V. Functional gastroduodenal disorders. Gastroenterology. 2006 Apr;130(5):1466-79. doi: 10.1053/j.gastro.2005.11.059. PMID 16678560
- [Result] Ford AC, Marwaha A, Lim A, Moayyedi P. What is the prevalence of clinically significant endoscopic findings in subjects with dyspepsia? Systematic review and meta-analysis. Clin Gastroenterol Hepatol. 2010 Oct;8(10):830-7, 837.e1-2. doi: 10.1016/j.cgh.2010.05.031. Epub 2010 Jun 10. PMID 20541625
- [Result] Olmos JI, Piskorz MM, Litwin N, Schaab S, Tevez A, Bravo-Velez G, Uehara T, Hashimoto H, Rey E, Sorda JA, Olmos JA. Exocrine Pancreatic Insufficiency is Undiagnosed in Some Patients with Diarrhea-Predominant Irritable Bowel Syndrome Using the Rome IV Criteria. Dig Dis Sci. 2022 Dec;67(12):5666-5675. doi: 10.1007/s10620-022-07568-8. Epub 2022 Jun 15. PMID 35704255